CLINICAL TRIAL: NCT02082353
Title: Analysis of Patients Treated for Chronic Granulomatous Disease Since January 1, 1995
Brief Title: Patients Treated for Chronic Granulomatous Disease (CGD) Since 1995
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rare Diseases Clinical Research Network (Network); Primary Immune Deficiency Treatment Consortium (PIDTC) (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT RDCRN PIDTC-6903; U54AI082973 (NIH)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Granulomatous Disease, Chronic
Keywords: Granulomatous Disease, Chronic; Hematopoietic Stem Cell Transplantation (HSCT); bone marrow transplant (BMT); non-transplant; factors associated with best outcomes of transplant in CGD
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood, skin swabs and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Retrospective CGD Cohort: Longitudinal analysis
- Prospective CGD Cohort: Longitudinal analysis
- HCT CGD Cohort: Cross-sectional analysis
- Conventional Non-Transplant CGD Cohort: Longitudinal analysis

SUMMARY:
Chronic granulomatous disease (CGD) is an inherited immune system abnormality in which bone marrow transplantation (BMT) has been shown to be curative. However the risks of transplantation are high and not all patients with CGD may need to undergo this high risk procedure. This study will determine the long term medical condition and daily functioning of participants with CGD after a transplant and if possible, compare these results to participants who do not undergo a transplant.

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is an immune deficiency where the neutrophils (a type of white blood cell that kills bacteria and fungi) do no work properly. Some individuals with CGD have neutrophils that do not work at all, whereas others have neutrophils that work partially, but not normally. In the past (over 20 years ago), most individuals with CGD were managed with antibiotics and antifungal medications alone. As the science of blood and marrow transplant (BMT) improved, some with CGD started to receive a BMT. It remained controversial whether individuals with CGD should receive a BMT or medical management alone (antibiotics, antifungals, and other treatments that do not include BMT).

The aim of this natural history study is to better define the role of BMT compared to medical management of CGD. Specifically, what are the outcomes of BMT versus medical management alone, why do some individuals with CGD benefit from BMT, and what are the long-term outcomes of both approaches. Researchers are interested in how individuals with CGD who have no neutrophil function may differ from those with some neutrophil function, how the types of infections and inflammatory complications of CGD impact on survival and how BMT may improve these complications. There are also questions as to how the types of bacteria (called the microbiome) found in the gastrointestinal tract (colon, large intestine) of individuals with CGD influences certain inflammatory complications (such as colitis), and how BMT changes the microbiome in individuals with CGD. All of this will help doctors in the future to better treat patients with CGD.

This study includes a retrospective (looking back into the past), cross-sectional (one time collection of information and/or research testing) and a prospective (looking from today and into the future) component. These are known as longitudinal studies (e.g., looking at information of participants over time).

Persons with CGD who were born 1988 to the present day are eligible, regardless of whether they received a BMT (as long as the BMT was after 1995) or medical therapy only. Individuals who are newly diagnosed with CGD can also be enrolled and followed longitudinally (over time), to determine their outcome from the choice of therapy that is made. An important component of this study is the 'cross sectional' study, where participants with more than 3 years of follow-up after transplant or diagnosis are asked to provide additional research blood work, and information is gathered regarding long-term transplant outcomes such as infections, graft-versus-host disease, autoimmune diseases, and quality of life. In addition, the participants will be asked to provide stool samples to allow investigators to look at how certain bacteria found in the gut (called the microbiome) affect complications of CGD, such as gastrointestinal disease. This will allow primary immune deficiency investigators/doctors to better understand the outcomes of different therapeutic approaches and to best design new treatments and clinical trials in the future for children with CGD.

ELIGIBILITY:
Inclusion Criteria:

* Participant Inclusion Criteria (Part 1 - Longitudinal Analysis)

  * CGD Patients Undergoing Transplant 1995 to Present with Birth Year In or After 1988

    1. CGD Patients will be Defined by both Defective Neutrophil NADPH Oxidase Function and by Clinical History Consistent with CGD

       Patients must have both of:

       A functional assay demonstrating abnormal NADPH oxidase function (see A below); AND Clinical history consistent with CGD (see B below).

       *************************************************************************

       Patients must have both "A" and "B":

       A. Function: Assays of NADPH Oxidase Function

       I. Dihydrorhodamine (DHR) Assay:
       * Blood sample was obtained at a time when patient was clinically stable and not critically ill, with control samples performed simultaneously indicating a qualified assay; and
       * Assay unequivocally demonstrates CGD with an stimulation index (SI) SI < 35 or equivalent. Assay report, including mean fluorescence intensity (MFI) from unstimulated and stimulated samples and gating strategy, must be de-identified and provided. OR

       II. Nitroblue Tetrazolium Oxidation Test (NBT):

       o Diagnostic of CGD (reported as reduced granulocyte oxidative response). Report must be de-identified and provided. AND

       B. Clinical History: One or More of the Following:
       * Severe and/or recurrent infection (liver, perirectal or lung abscess; pneumonia; adenitis; or osteomyelitis) due to, for example, Staphylococcus aureus, Burkholderia sp, Serratia marcescens, non-albicans Candida sp, Aspergillus sp or other mold; or Nocardia sp or other deep tissue infection characteristic of CGD
       * Sterile granulomatous disease in respiratory, gastrointestinal or urogenital tracts; or Crohn's disease-like colitis
       * A family history consistent with either X-linked or autosomal recessive CGD

       In cases where either functional assay (A) or history (B) is equivocal, one or more of the following may be used to confirm a diagnosis of CGD:

       C. Absent or significantly reduced in expression or abnormal size of any of the 5 phox components (gp91 phox, p47 phox, p22 phox, p67phox, and p40phox) of NADPH oxidase, by either:
       * Western blot
       * Northern blot OR D. Mutation in a gene encoding one of the 5 phox components (gp91 phox, p47 phox, p22 phox, p67 phox, and p40 phox) of NADPH oxidase that is predictive of a decreased or absent oxidative burst. (Nonsense, frameshift, or previously described missense mutation associated with CGD).

       Molecular Diagnosis is Desirable In addition, molecular diagnosis (gene sequencing and expression analysis) of CGD is desirable and should be performed when possible.
    2. Further Characterization of Oxidase Level, Longitudinal Study, Prospective Cohort Patients who are to undergo transplantation during the study period must be further characterized as oxidase-null or oxidase positive by level of oxidase production by either:

       * DHR assay stimulation Index: where SI ≤ 2.5 will be classified as oxidase-null CGD. Those with SI > 2.5 will be classified as oxidase positive CGD. A single validated test that is accepted by the PID-CGD Review Panel is adequate, but testing on two occasions for validation is desirable. OR
       * Ferricytochrome C reduction assay of granulocytes with O2 < 2.3 nmoles /106 cells/h classified as oxidase-null CGD. A single validated test that is accepted by the PID-CGD Review Panel is adequate, but testing on two occasions for validation is desirable.

       OR

       o Genetic sequencing reporting a mutation that is unequivocally associated to absent oxidase production. (e.g. null mutations) will be classified as oxidase-null CGD (See discussion in Appendix I for how family history, genotype and CGD mutation information will be applied to assigning patients lacking any quantitative oxidase activity measurements to residual oxidase-null or residual oxidase-positive groups).
    3. Longitudinal Study, Retrospective Cohort Patients who have already been transplanted will be included regardless of whether further characterization by oxidase level (or genotype/mutation data) is possible or not.
  * Non-Transplanted CGD Patients with Birth Year In or After 1988 A non-transplant (conventional therapy) group of CGD subjects will be enrolled in the longitudinal study. The non-transplant subjects will be selected from the potentially eligible (retrospective) patient cohort with diagnosis of CGD treated with conventional non-transplant therapy. Participating sites will enter their entire retrospective cohort of CGD patients having birth year in or after 1988 into the registration cohort for this protocol. Baseline for both non-transplant subjects and HCT subjects for the purpose of comparing survival will be the year of birth. However, for non-transplant subjects, many of the detailed analyses such as infection and autoimmune complication rates will be assessed in the year preceding the date of last contact.
* Participant Inclusion Criteria (Part 2 - Cross-Sectional Analysis) To participate in the Cross-Sectional Analysis, patients must have previously been enrolled into the Longitudinal Analysis of Protocol 6903. All transplanted subjects in the Cross-Sectional Analysis are surviving and shall have at least 3 years of follow-up post-transplant to be included. Non-transplanted CGD subjects will become eligible for consideration for the Cross-Sectional Analysis if they were eligible and enrolled in the retrospective cohort of the Longitudinal Analysis, and if/when they are > 3 years post-diagnosis of CGD. Provision of written informed consent will be required for inclusion in the Cross-Sectional Analysis.

Exclusion Criteria:

* Participant Exclusion Criteria (Longitudinal and Cross- Sectional Analyses)

  * Presence of other primary immunodeficiency syndromes that do not meet the clinical and laboratory criteria for CGD.
  * Rac2 Deficiency
  * Myeloperoxidase Deficiency (MPO Deficiency)
  * Glutathione deficiency
  * Leukocyte adhesion deficiency syndrome
* Non-transplant subjects:

  * The above exclusions pertain.
  * In addition, non-transplant subjects will be excluded if the only assessment of oxidase function available is the nitroblue tetrazolium (NBT) test (a non-quantitative test).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Institutions participating in Rare Diseases Clinical Research Network (RDCRN)
Sampling Method: Non-Probability Sample
Enrollment: 1480 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Death | HCT to date of death, up to an expected average of 3 years
  The event analyzed is death from any cause. The time from HCT to death or last follow up will be analyzed. Cause of death will also be collected. Surviving patients will be censored at the time of last observation.

SECONDARY OUTCOMES:
Engraftment | an expected average of 3 years
  Engraftment will be measures in whole blood using either fluorescent in situ hybridization (FISH) for sex chromosomes or short tandem repeat polymerase chain reaction (PCR) or (STRs) in whole blood.
Quality of Life Measures | an expected average of 3 years
  Age appropriate testing will be performed at the cross-sectional visit in patients surviving at least two years posttransplant:
  * Pediatrics quality of life (QL) Family Impact Module, Parent Report
  * Peds QL Infant Scales Module (ages 1-24 months), Parent Report
  * Peds QL Generic Core Scales for Toddlers (ages 2-4 yr), Parent Report
  * Peds QL Generic Core Scales (ages 5-25 yr), Child/Parent Reports
  * Peds QL Transplant Module
  * Standard Form (SF)-36 (adult)
  * Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT BMT) (adult)
Infections | an expected average of 3 years
  CGD or transplant-related and transplant-related infection
Autoimmune or inflammatory complications | an expected average of 3 years
  - For HCT subjects, inflammation (inflammatory complications) includes chronic graft-versus-host disease (GVHD)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Puck, MD, Principal Investigator — University of California, San Francisco; Donald B. Kohn, MD, Principal Investigator — University of California, Los Angeles
Locations (44):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA, Los Angeles, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California (UCSF) Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. duPont Hospital for Children/Nemours, Wilmington, Delaware
  - Children's National Medical Center, Washington DC, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital - St. Petersburg, FL, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of New Orleans at LSUHSC, New Orleans, Louisiana
  - NIH Clinical Center Genetic Immunotherapy Section, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Cardinal Glennon Children's Hospital/ St. Louis University, St Louis, Missouri
  - Washington University/ St.Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-kettering Cancer Center, New York, New York
  - University of Rochester Medical Center/ Golisano Children's Hospital, Rochester, New York
  - New York Medical College, Maria Fareri Children's Hospital, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies/ University Hospitals Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Methodist Children's Hospital of South Texas/Texas Transplant Institute, San Antonio, Texas
  - Primary Children's Medical Center/ University of Utah, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle, Washington
  - University of Wisconsin/ American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin-Milwaukee, Milwaukee, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU St. Justine, Montreal, Quebec

REFERENCES:
- [Background] Griffith LM, Cowan MJ, Kohn DB, Notarangelo LD, Puck JM, Schultz KR, Buckley RH, Eapen M, Kamani NR, O'Reilly RJ, Parkman R, Roifman CM, Sullivan KE, Filipovich AH, Fleisher TA, Shearer WT. Allogeneic hematopoietic cell transplantation for primary immune deficiency diseases: current status and critical needs. J Allergy Clin Immunol. 2008 Dec;122(6):1087-96. doi: 10.1016/j.jaci.2008.09.045. Epub 2008 Nov 6. PMID 18992926
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Pai SY, Ballard B, Bauer SC, Bleesing JJ, Boyle M, Brower A, Buckley RH, van der Burg M, Burroughs LM, Candotti F, Cant AJ, Chatila T, Cunningham-Rundles C, Dinauer MC, Dvorak CC, Filipovich AH, Fleisher TA, Bobby Gaspar H, Gungor T, Haddad E, Hovermale E, Huang F, Hurley A, Hurley M, Iyengar S, Kang EM, Logan BR, Long-Boyle JR, Malech HL, McGhee SA, Modell F, Modell V, Ochs HD, O'Reilly RJ, Parkman R, Rawlings DJ, Routes JM, Shearer WT, Small TN, Smith H, Sullivan KE, Szabolcs P, Thrasher A, Torgerson TR, Veys P, Weinberg K, Zuniga-Pflucker JC; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) report. J Allergy Clin Immunol. 2014 Feb;133(2):335-47. doi: 10.1016/j.jaci.2013.07.052. Epub 2013 Oct 15. PMID 24139498
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Shearer WT, Burroughs LM, Torgerson TR, Decaluwe H, Haddad E; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) update. J Allergy Clin Immunol. 2016 Aug;138(2):375-85. doi: 10.1016/j.jaci.2016.01.051. Epub 2016 Apr 22. PMID 27262745
- [Result] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Result] Haddad E, Allakhverdi Z, Griffith LM, Cowan MJ, Notarangelo LD. Survey on retransplantation criteria for patients with severe combined immunodeficiency. J Allergy Clin Immunol. 2014 Feb;133(2):597-9. doi: 10.1016/j.jaci.2013.10.022. Epub 2013 Dec 10. No abstract available. PMID 24331379
- [Result] Shearer WT, Dunn E, Notarangelo LD, Dvorak CC, Puck JM, Logan BR, Griffith LM, Kohn DB, O'Reilly RJ, Fleisher TA, Pai SY, Martinez CA, Buckley RH, Cowan MJ. Establishing diagnostic criteria for severe combined immunodeficiency disease (SCID), leaky SCID, and Omenn syndrome: the Primary Immune Deficiency Treatment Consortium experience. J Allergy Clin Immunol. 2014 Apr;133(4):1092-8. doi: 10.1016/j.jaci.2013.09.044. Epub 2013 Nov 28. PMID 24290292
- [Result] Dvorak CC, Cowan MJ, Logan BR, Notarangelo LD, Griffith LM, Puck JM, Kohn DB, Shearer WT, O'Reilly RJ, Fleisher TA, Pai SY, Hanson IC, Pulsipher MA, Fuleihan R, Filipovich A, Goldman F, Kapoor N, Small T, Smith A, Chan KW, Cuvelier G, Heimall J, Knutsen A, Loechelt B, Moore T, Buckley RH. The natural history of children with severe combined immunodeficiency: baseline features of the first fifty patients of the primary immune deficiency treatment consortium prospective study 6901. J Clin Immunol. 2013 Oct;33(7):1156-64. doi: 10.1007/s10875-013-9917-y. Epub 2013 Jul 2. PMID 23818196
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Puck JM, Buckley RH, Candotti F, Conley ME, Fleisher TA, Gaspar HB, Kohn DB, Ochs HD, O'Reilly RJ, Rizzo JD, Roifman CM, Small TN, Shearer WT; Workshop Participants. Improving cellular therapy for primary immune deficiency diseases: recognition, diagnosis, and management. J Allergy Clin Immunol. 2009 Dec;124(6):1152-60.e12. doi: 10.1016/j.jaci.2009.10.022. PMID 20004776
- [Result] Marsh RA, Leiding JW, Logan BR, Griffith LM, Arnold DE, Haddad E, Falcone EL, Yin Z, Patel K, Arbuckle E, Bleesing JJ, Sullivan KE, Heimall J, Burroughs LM, Skoda-Smith S, Chandrakasan S, Yu LC, Oshrine BR, Cuvelier GDE, Thakar MS, Chen K, Teira P, Shenoy S, Phelan R, Forbes LR, Chellapandian D, Davila Saldana BJ, Shah AJ, Weinacht KG, Joshi A, Boulad F, Quigg TC, Dvorak CC, Grossman D, Torgerson T, Graham P, Prasad V, Knutsen A, Chong H, Miller H, de la Morena MT, DeSantes K, Cowan MJ, Notarangelo LD, Kohn DB, Stenger E, Pai SY, Routes JM, Puck JM, Kapoor N, Pulsipher MA, Malech HL, Parikh S, Kang EM; submitted on behalf of the Primary Immune Deficiency Treatment Consortium. Chronic Granulomatous Disease-Associated IBD Resolves and Does Not Adversely Impact Survival Following Allogeneic HCT. J Clin Immunol. 2019 Oct;39(7):653-667. doi: 10.1007/s10875-019-00659-8. Epub 2019 Aug 2. PMID 31376032
- [Derived] Chandrasekaran P, Han Y, Zerbe CS, Heller T, DeRavin SS, Kreuzberg SA, Marciano BE, Siu Y, Jones DR, Abraham RS, Stephens MC, Tsou AM, Snapper S, Conlan S, Subramanian P, Quinones M, Grou C, Calderon V, Deming C, Leiding JW, Arnold DE, Logan BR, Griffith LM, Petrovic A, Mousallem TI, Kapoor N, Heimall JR, Barnum JL, Kapadia M, Wright N, Rayes A, Chandra S, Broglie LA, Chellapandian D, Deal CL, Grunebaum E, Lim SS, Mallhi K, Marsh RA, Murguia-Favela L, Parikh S, Touzot F, Cowan MJ, Dvorak CC, Haddad E, Kohn DB, Notarangelo LD, Pai SY, Puck JM, Pulsipher MA, Torgerson TR, Kang EM, Malech HL, Segre JA, Bryant CE, Holland SM, Falcone EL. Intestinal microbiome and metabolome signatures in patients with chronic granulomatous disease. J Allergy Clin Immunol. 2023 Dec;152(6):1619-1633.e11. doi: 10.1016/j.jaci.2023.07.022. Epub 2023 Sep 1. PMID 37659505
- [Derived] Leiding JW, Arnold DE, Parikh S, Logan B, Marsh RA, Griffith LM, Wu R, Kidd S, Mallhi K, Chellapandian D, Si Lim SJ, Grunebaum E, Falcone EL, Murguia-Favela L, Grossman D, Prasad VK, Heimall JR, Touzot F, Burroughs LM, Bleesing J, Kapoor N, Dara J, Williams O, Kapadia M, Oshrine BR, Bednarski JJ, Rayes A, Chong H, Cuvelier GDE, Forbes Satter LR, Martinez C, Vander Lugt MT, Yu LC, Chandrakasan S, Joshi A, Prockop SE, Davila Saldana BJ, Aquino V, Broglie LA, Ebens CL, Madden LM, DeSantes K, Milner J, Rangarajan HG, Shah AJ, Gillio AP, Knutsen AP, Miller HK, Moore TB, Graham P, Bauchat A, Bunin NJ, Teira P, Petrovic A, Chandra S, Abdel-Azim H, Dorsey MJ, Birbrayer O, Cowan MJ, Dvorak CC, Haddad E, Kohn DB, Notarangelo LD, Pai SY, Puck JM, Pulsipher MA, Torgerson TR, Malech HL, Kang EM. Genotype, oxidase status, and preceding infection or autoinflammation do not affect allogeneic HCT outcomes for CGD. Blood. 2023 Dec 14;142(24):2105-2118. doi: 10.1182/blood.2022019586. PMID 37562003
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: Primary Immune Deficiency Treatment Consortium (PIDTC) — https://www.rarediseasesnetwork.org/spotlight/v9i1/PIDTC
- See also: Rare Diseases Clinical Research Network — https://www.rarediseasesnetwork.org/research-groups